CLINICAL TRIAL: NCT05900297
Title: Antibiotic Regimen for Patients Seeking Dental Implants Procedures
Brief Title: Antibiotic Regimen for Dental Implants Cases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Salma Mohamed Essam El-din Osman, medical doctor, Assiut University
Other Study IDs: antibiotic for dental implants
Record Dates: First submitted 2023-05-27; First posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Dental Implant Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to:

1. To identify the most common organisms causing dental implant failure.
2. Set an appropriate antibiotic regimen according to the causative organism to limit the antimicrobial resistance by limit the use of antibiotics.

DETAILED DESCRIPTION:
Dental implant surgery is a common treatment for replacing missing teeth and has a high success rate. Implant failure is most likely the result of multiple factors as Age, sex, smoking, maxillary implant site, quantity and quality of bone, implant surface treatments and features are some of the statistically examined parameters linked to implant failure. The most frequent and avoidable cause of dental implant failure is infection. A retrospective analysis demonstrated fewer numbers of early implant failures among those that were placed under antibiotic treatments.

Early implant failure is commonly associated with certain strains of bacteria. The most common bacteria involved are streptococci, anaerobic Gram-positive cocci, and anaerobic Gram-negative rods.Porphyromonas gingivalis and Fusobacterium nucleatum frequently colonize the implant in early and late losses and could therefore be characteristic for implant loss in general.

Thus, the antibiotic to prevent delayed healing of wound should be bactericidal and of low toxicity. Systemic antibiotic prophylaxis has been used to reduce the risk of early implant failure and local infections around dental implants.Antibiotics are one of the most cost-effective, life-saving medicines and contribute to an extended lifespan. Access to antibiotics without a prescription is a driving factor for irrational antibiotic use due to a potential lack of access to proper diagnosis and diagnostic tools. This eventually leads to the development and spread of antibiotic resistance &it is one of the increasing public health challenges worldwide.

ELIGIBILITY:
Inclusion Criteria: Saliva samples from patients seeking dental implant procedures

-

Exclusion Criteria:

* Immunodeficiency or immunosuppressing treatment
* current antibiotic treatment
* smoking
* acute or chronic oral infection (including ongoing periodontal infection).

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients seeking dental implant procedures
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-15 (Estimated); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-20 (Estimated)

PRIMARY OUTCOMES:
to limit the antimicrobial resistance by identifying the most suitable antibiotic regimen according to the intra-oral organisms | september 2023-september 2024
  according to the antibiogram at least 30 isolates from each species are needed to identify the most common organisms and set an appropriate antibiotic regimen for patients seeking dental implants.An antibiogram is an overall profile of antimicrobial susceptibility testing results of a specific microorganism to a battery of antimicrobial drugs. This profile is generated by the laboratory using aggregate data from a hospital or healthcare system; data are summarized periodically and presented showing percentages of organisms tested that are susceptible to a particular antimicrobial drug

SECONDARY OUTCOMES:
to prevent dental implant failure by setting the most suitable antibiotic regimen according to the intra-oral micro-organisms | through the study completion, an average of one year.
  the investigator can define and set antibiotic regimen to the oral micro-organisms by the antibiogram .The Clinical and Laboratory Standards Institute (CLSI; formerly NCCLS) published guidelines entitled "Analysis and Presentation of Cumulative Antimicrobial Susceptibility Test Data" for use when creating an antibiogram. CLSI guidelines recommend compiling the antibiogram at least annually, including only the first isolate per patient in the period analyzed, and including only organisms for which ≥30 isolates were tested in the period analyzed.

REFERENCES:
- [Background] Kochar SP, Reche A, Paul P. The Etiology and Management of Dental Implant Failure: A Review. Cureus. 2022 Oct 19;14(10):e30455. doi: 10.7759/cureus.30455. eCollection 2022 Oct. PMID 36415394
- [Background] Surapaneni H, Yalamanchili PS, Basha MH, Potluri S, Elisetti N, Kiran Kumar MV. Antibiotics in dental implants: A review of literature. J Pharm Bioallied Sci. 2016 Oct;8(Suppl 1):S28-S31. doi: 10.4103/0975-7406.191961. PMID 27829741
- [Background] Machowska A, Stalsby Lundborg C. Drivers of Irrational Use of Antibiotics in Europe. Int J Environ Res Public Health. 2018 Dec 23;16(1):27. doi: 10.3390/ijerph16010027. PMID 30583571
- [Background] Momand P, Becktor JP, Naimi-Akbar A, Tobin G, Gotrick B. Effect of antibiotic prophylaxis in dental implant surgery: A multicenter placebo-controlled double-blinded randomized clinical trial. Clin Implant Dent Relat Res. 2022 Feb;24(1):116-124. doi: 10.1111/cid.13068. Epub 2022 Jan 24. PMID 35075765
- [Background] Korsch M, Marten SM, Stoll D, Prechtl C, Dotsch A. Microbiological findings in early and late implant loss: an observational clinical case-controlled study. BMC Oral Health. 2021 Mar 11;21(1):112. doi: 10.1186/s12903-021-01439-w. PMID 33706748
- [Background] Bernabeu-Mira JC, Penarrocha-Diago M, Penarrocha-Oltra D. Prescription of Antibiotic Prophylaxis for Dental Implant Surgery in Healthy Patients: A Systematic Review of Survey-Based Studies. Front Pharmacol. 2021 Feb 10;11:588333. doi: 10.3389/fphar.2020.588333. eCollection 2020. PMID 33643035
- [Background] Antwi AN, Stewart A, Crosbie M. Fighting antibiotic resistance: a narrative review of public knowledge, attitudes, and perceptions of antibiotics use. Perspect Public Health. 2020 Nov;140(6):338-350. doi: 10.1177/1757913920921209. Epub 2020 Jun 9. PMID 32515278
- [Background] Pyysalo M, Helminen M, Antalainen AK, Sandor GK, Wolff J. Antibiotic prophylaxis patterns of Finnish dentists performing dental implant surgery. Acta Odontol Scand. 2014 Nov;72(8):806-10. doi: 10.3109/00016357.2014.913194. Epub 2014 May 5. PMID 24791607
- [Background] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627